CLINICAL TRIAL: NCT06668077
Title: Inhibitory Control Training and Theta Burst Transcranial Magnetic Stimulation (iTBS) for Treating People With Excess Weight: Behavioral and Brain Changes (InhibE).
Brief Title: Inhibitory Control Training and iTBS for Excess Weight: Behavioral and Brain Changes (InhibE).
Acronym: InhibE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raquel Vilar López (Other)
Collaborators: Government of Spain (Unknown)
Responsible Party: Sponsor-Investigator, Raquel Vilar López, Principal Investigator, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SICEIA-2024-000656
Record Dates: First submitted 2024-09-30; First posted 2024-10-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Overweight and Obesity; Inhibition, Psychological
Keywords: excess weight; overweight; inhibitory control; cognitive training; iTBS
MeSH Terms: conditions — Overweight; Obesity; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The psychologists that conduct the assessments (screening, assessment sessions and follow-ups) will be blinded to the group allocation during the whole project. Further, all participants will be blind to their condition. Also, the people who perform the statistical analyses will be blind to the condition of the groups, through the coding of the interventions. Only the therapist performing the interventions will not be blind to the allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined intervention (Experimental): Experimental: Active iTBS of the DLPFC combined with inhibitory control training. An experimental group will receive: i) an informative session; ii) 4 pre treatment sessions (one assessment session with questionnaires, one with fMRI and one with biological samples. Also, a counselling session on diet and on physical exercise); iii) participate in 2 weekly individual intervention sessions that consist of iTBS of the left DLPFC (10 min) followed immediately by inhibitory control training for 10 minutes; iv) 3 sessions of post treatment assessment (one with questionnaires, one with fMRI and one with biological samples); v) 2 follow-up assessment sessions (3 months after completing the intervention) to repeat questionnaires and biological samples
  Interventions: Device: iTBS of the left DLPFC; Behavioral: Inhibitory control training
- Active iTBS (Active Comparator): Experimental: Active iTBS of the DLPFC only. An experimental group will receive: i) an informative session; ii) 4 pre treatment sessions (one assessment session with questionnaires, one with fMRI and one with biological samples. Also, a counselling session on diet and on physical exercise); iii) participate in 2 weekly individual intervention sessions that consist of iTBS of the left DLPFC that will last about 10 minutes each; iv) 3 sessions of post treatment assessment (one with questionnaires, one with fMRI and one with biological samples); v) 2 follow-up assessment sessions (3 months after completing the intervention) to repeat questionnaires and biological samples
  Interventions: Device: iTBS of the left DLPFC
- Sham iTBS (Sham Comparator): Control: iTBS of the vertex (sham). The control group will receive: i) an informative session; ii) 4 pre treatment sessions (one assessment session with questionnaires, one with fMRI and one with biological samples. Also, a counselling session on diet and on physical exercise); iii) participate in 2 weekly individual intervention sessions that consist of iTBS of the vertex that will last about 10 minutes each; iv) 3 sessions of post treatment assessment (one with questionnaires, one with fMRI and one with biological samples); v) 2 follow-up assessment sessions (3 months after completing the intervention) to repeat questionnaires and biological samples
  Interventions: Device: iTBS of the vertex

INTERVENTIONS:
Device: iTBS of the left DLPFC — Participants will receive a 3 minutes active theta burst transcranial magnetic stimulation (iTBS) of the DLPFC of the left hemisphere while not performing any other task
  Other Names: Active iTBS
  Arms: Active iTBS; Combined intervention
Device: iTBS of the vertex — Participants will receive a 3 minutes active theta burst transcranial magnetic stimulation (iTBS) of the vertex while not performing any other task
  Other Names: Sham iTBS
  Arms: Sham iTBS
Behavioral: Inhibitory control training — Computerized cognitive training. Participants will perform the task of the FoodT app for 10 minutes during two weeks (taking advantage of time of maximum brain potentiation after the iTBS, Rossi et al., 2009). Images of food and non-food appear on the left, right or centre of the smart phone screen and participants must touch it (or not, depending on the cue) with their index finger as quickly as possible. Participants earn points for correct tap responses and lose points for incorrect tap responses. If the image has a green border around it, participants must tap the image and win 1 point. But if the image has a red border around it, participants must inhibit the tapping response, otherwise 1 point will be lost. Participants must respond as quickly and accurately as possible. Pictures of healthy and unhealthy foods are always paired with the Go and the No-Go signal, respectively. Non-food images are paired 50% of the time with the Go and the No-Go signal
  Other Names: FoodT
  Arms: Combined intervention

SUMMARY:
People with excess weight (EW) are characterized by high impulsivity, high levels of craving for high-calorie foods, deficits in inhibitory control, and maladaptive decision-making. These characteristics are related, at the brain level, to alterations in the activation of areas such as the dorsolateral prefrontal cortex (DLPFC) and its connectivity. The proposed intervention seeks to target these issues. Thus, the present study aims to characterize the effects of neuromodulation with intermittent theta burst transcranial magnetic stimulation (iTBS) of the DLPFC alone and in combination with inhibitory control training to produce brain, cognitive and behavioral changes, and modify altered biological parameters in people with EW. Participants will be randomly allocated to one of three groups: (1) a group that will receive active iTBS of the DLPFC combined with inhibitory control training with a food Go/No-go paradigm, (2) a group that will receive active iTBS of the DLPFC only, and (3) a control group that will receive sham iTBS. It is hypothesized that the combined intervention will obtain better results that the neuromodulation alone, and that both interventions, compared to sham iTBS, will achieve: (i) decreased body mass index, (ii) decreased craving, (iii) modified brain connectivity and activation both at rest and linked to task performance with food stimuli, (iv) improved anthropometric measures (waist circumference and waist-to-hip and waist-to-height ratios), (v) improved eating and exercise behaviors (decreased caloric intake and increased frequency and time of physical activity), (vi) improved emotional symptoms and emotional eating (depression, anxiety, emotional regulation, emotional eating, reward-related eating, non-homeostatic eating), (vii) improved cognitive abilities (motor and cognitive inhibition, delay of gratification, impulsivity, working memory, cognitive flexibility and decision making), (viii) changes in biological parameters associated to the interventions (plasma and microbiota), and (ix) advantages in cost-effectiveness and cost-utility based on economic evaluation analyses.

DETAILED DESCRIPTION:
1. STARTING HYPOTHESES AND GENERAL OBJECTIVE HYPOTHESIS:

   HYPOTHESIS: Neuromodulation with iTBS applied to the left DLPFC in combination with inhibitory control training with a food Go/No-go paradigm will be associated with decreased (i) BMI, and (ii) craving; (iii) modified brain connectivity and activation both at rest and linked to task performance with food stimuli; improved (iv) anthropometric measures (waist circumference and waist-to-hip and waist-to-height ratios), (v) eating and exercise behaviors (caloric intake increased frequency and time of physical activity), (vi) emotional symptoms and emotional eating (depression, anxiety, emotional regulation, emotional eating, reward-related eating, non-homeostatic eating), (vii) cognitive abilities (motor and cognitive inhibition, delay of gratification, impulsivity, working memory, cognitive flexibility and decision making); (viii) changes in biological parameters (plasma and microbiota), and (ix) advantages in cost-effectiveness and cost-utility based on economic evaluation analyses.

   GENERAL OBJECTIVE: To determine the effects of neuromodulation with iTBS in DLPFC alone and in combination with inhibitory control training to generate brain, behavioural, emotional, cognitive and biological changes in people with EW.

   1.1. Specific Aims: Objective 1: To determine the effectiveness of iTBS of the DLPFC as an add-on to the treatment as usual (TAU: diet and exercise) for the treatment of people with excess weight (improvements in BMI, craving, anthropometric measures, food and exercise behaviours, emotional symptoms and emotional eating, cognitive measures and biological parameters).

   Objective 2: To study the effectiveness of combining iTBS and inhibitory control training compared to iTBS alone (both as an add-on to TAU), for the treatment of EW (using the same parameters before) Objective 3: To characterize the effects of neuromodulation with iTBS of DLPFC alone and in combination with inhibitory control training to modify brain connectivity and activation both at rest and linked to task performance with food stimuli with functional magnetic resonance imaging (fMRI).

   Objective 4: To determine the relationship of biological parameters obtained in blood, saliva, urine and faeces, as well as candidate genes, with neuropsychological variables (depression, anxiety, stress, emotional regulation, emotional eating, craving, motor and cognitive inhibition, food valuation, delay of gratification, impulsivity, working memory, flexibility and decision making) and brain neuroimaging (activation, grey and white matter volume and connectivity).

   Objective 5: To analyse the economic evaluation of the cost-effectiveness and cost-utility of combined training (neuromodulation with iTBS and inhibitory control training) in people with EW, and to analyse the budgetary impact of the program if it were to be implemented in the national health system.
2. METHODOLOGY 2.1. Design: Randomized controlled trial of parallel groups. 2.2. Sample size and statistical power: The sample size was calculated using the G*Power 3.1 tool G-Power v3.1.9.7. To do so, we relied on the only study to date that has analysed changes in BMI in people with obesity after the administration of 4 rTMS sessions over 2 weeks, which found a small effect size (Cohen's d= 0.31). Thus, considering a small effect size for conducting ANOVAs (f= 0.15), the minimum recommended sample size to reach a power of 0.95 and alpha level of 0.05 to calculate the interaction model of the three groups (combined intervention vs. neuromodulation alone vs. sham iTBS) and three repeated measures was 141 (47 participants per group).

   Pre-treatment sessions: information, dietary plus physical guidelines (all groups):

   All participants will participate in a group briefing informational session about the procedure and rationale of the study that will last about an hour. Also, informative videos and brochures will be provided. After that, there will be two 90-minute sessions given by a nutritionist and personal trainer respectively to provide individualized diet and physical exercise instructions.

   Neurocognitive intervention:

   Duration: 2 weeks of 5 daily sessions. Part 1 (all groups). Three minutes of neuromodulation with iTBS (in the DLPFC for groups 1 and 2; in the vertex for group 3). The whole process of iTBS includes 3 minutes of stimulation and time devoted to coil location, reception and farewell (10 minutes).

   Part 2 (group 1). Immediately after the iTBS, only group 1 will also receive a 10-minute inhibition training with the FoodT app in their smart phones.

   In this task, participants are instructed to touch green circled items as quickly as possible, but to withhold their response and not to press on the red circled items. Some images are food (high-calorie and low-calorie), some non-foods. Participants can choose which food categories would like to train to resist, and those high-calorie foods are always paired with the no-go signal.
3. PROCEDURE Assessments will be delivered online through LimeSurvey and Milliseconds platforms. Inclusion and exclusion criteria will be checked.

All candidates who meet the criteria will attend an information meeting to receive written and oral information about the project and will be asked for their informed consent. Then, participants will be randomly assigned to groups before the pre-treatment assessment sessions. A simple randomization will be performed by generating five-letter codes with Calculado.net and randomizing the codes into three different groups using Rafflys. The three groups of the study will complete three assessments (pre, post, 3-month follow-up). What will differentiate the groups will be, therefore, the treatment: iTBS applied to the DLPFC followed by inhibitory control training vs. iTBS applied to the DLPFC vs. iTBS applied to the vertex (sham). At the end of the project, if an intervention is effective, the other groups will be offered the possibility of receiving it.

Informative and evaluation sessions will be developed in groups of 4-6 people. iTBS sessions will be administered individually. If a participant misses a session, it will be rescheduled for the beginning of the next week at a similar time. There will be at least 8 experimental groups of DLPFC neuromodulation combined with inhibitory control training (45 participants), 8 experimental groups of DLPFC neuromodulation alone (45 participants) and 8 control groups of sham iTBS (45 participants). The program will comprise 6 weeks including: three assessments (pre, post, and 3-month follow-up), ten intervention sessions (two weeks of 5 daily sessions), information and the diet and exercise sessions too. Assessment sessions will last about 2 hours while intervention sessions will between 10 and 20 minutes depending on the group. The contents of each of the sessions will be as follows:

1. Informative session (session 1; week 1): For the participants to understand the foundation of the intervention information about the aims, basis of the project and the procedure of the research will be given. Participants will be provided written informed consent as well. At the end of this session, participants will be asked for their informed written consent.
2. Pre-treatment assessment (session 2, 3 and 4; week 2): All participants will complete, in session 2, the following instruments to assess the main and secondary outcomes, and the exploratory and economic measures: WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, CFA, IPAQ, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36, SOCRATES 00, QEWP-5, sociodemographic questionnaire, another one about used health resources, stigma and previous treatments questions. Also, all participants will undergo the fMRI session (session 3) and biological sample collection (blood, saliva, feces and urine) and anthropometric measures to calculate BMI, WC, WHR and WHtR (session 4).
3. Nutrition and physical exercise session (session 5; week 3): Participants will receive information on healthy nutritional (Ph.D. Nutritionist) and physical exercise (Ph.D. Sports Science) habits. In addition, participants will receive individualized diet and physical exercise guidelines, and participants will be able to consult any doubts to both professionals through WhatsApp groups.
4. Intervention sessions (sessions 6 to 15; weeks 4 and 5): Intervention will consist of five weekly individual sessions for two weeks, with a 10-20-minute total duration each. The stimulation parameters are based on the protocols for the application of iTBS in people with food intake problems, by Barone et al., (2023), and following international safety recommendations. The procedure in the three groups consists of:

   A. Localization of the stimulation area by T1 sequence structural neuroimaging images using the Brainsight software for the correct placement of the stimulation coil: in the active stimulation group it will be the left DLPFC area (x -37, y -34, z 78) corresponding to F3 position on the 10-20 EEG system. In the control group it will be the vertex (x 0, y-34, z 78), an area without cognitive effects after stimulation but matching the sensory effects.

   B. Neuromodulation applying an intermittent TBS with Megastim Rapid 2 magnetic stimulator and figure-8-coil: iTBS for 3 minutes with parameters of frequency 50 Hz, number of pulses 3; number of bursts 10; cycle duration 8 seconds; number of cycles 20; burst frequency 5 Hz; and total number of pulses 600. The stimulation intensity will be maintained at 30% of the stimulator's maximum output.

   C. Cognitive inhibitory control training (10 minutes): It will be performed with the FoodT app, for 10 minutes and will be applied immediately after the iTBS, taking advantage of its time of maximum brain potentiation. In this app, the task consists of touching as quickly as possible the items that appear surrounded with a green circle, and not responding to the items surrounded by a red circle. Some images correspond to food and others are not related to food. Participants can select the categories of the images to train, which should correspond to the foods used for binge eating (candy/gummies, cakes, chocolate, cookies, alcohol, chips, bread, cheese, fast food - burgers, take-out food -, sweet sodas, meat, pizza). Inhibitory control training consists of pairing high-calorie foods with the no-go signal.
5. Post-treatment assessment (session 16; week 6): To evaluate the effectiveness of the interventions, BMI and craving (FCQ-T/S-r) will be registered (main outcomes), and the following instruments will be administered to obtain the secondary outcomes; WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, CFA, IPAQ, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36 and a questionnaire about used health resources. Also, fMRI and biological samples of the pre-treatment assessment will be repeated.
6. Follow-up assessment (sessions 17; week 18): Follow-up at 3 months after the intervention will include the following measures: WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, CFA, IPAQ, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36, sociodemographic questionnaire and another one about used health resources, and collection of biological samples and anthropometric measures to obtain the main and secondary outcome measures.

Participants will be instructed to eat two hours before assessments (pre- and post-treatment, and the follow-up) and iTBS sessions. All the assessments will be carried out at the same hour.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 39.9
* Age between 18 and 60 years
* Proficiency in the Spanish language
* Right lateral dominance to avoid differential effects due to cortical hemispheric specialization

Exclusion Criteria:

* Traumatic, digestive, metabolic or systemic disorders that affect the central nervous system, autonomic or endocrine
* Severe psychopathological disorders and suicidal ideation or treatment for depression
* Eating disorders
* Contraindication for performing fMRI (pregnancy, metal implants, etc.) or iTBS (tinnitus, dizziness, surgical interventions, diseases or drugs that affect the CNS, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Change in BMI: Weight and height will be combined to report BMI in kg/m^2. Weight will be obtained in kilograms with a digital scale (TANITA Corporation of America) and height in meters with a measuring rod (SECA Tape Measure 206).
Changes in brain activation during a inhibitory control task (neuroimaging measures) | Pre-treatment assessment (week 2) and post-treatment assessment (week 6)
  Food Go/No-go task (Based on the FoodTrainer App; Lawrence et al., 2015): Pictures appear and afterwards a green (Go signal) or red (No-Go signal) circle appears around them. Participants are instructed to score points by answering with a knob if the image is surrounded by a green circle, but not to press when the image is surrounded by a red circle. The presentation of the images is the same as in the FoodTrainer application: 50% of the images are food, with 100% of the healthy ones being presented under the 'Go' condition and 100% of the unhealthy ones under the 'No-Go' condition. The remaining 50% are non-food images, with 50-50% paired with 'Go' and 'No-Go' cues. In addition, participants can choose which categories of unhealthy foods they want to train. Brain activation to Go vs. No-Go stimuli and food vs. non-food stimuli will be compared. The task will be analysed to assess the brain activity associated with the task, using a psychophysiological interaction analysis(PPI).

SECONDARY OUTCOMES:
Changes in Food decision-making (neuroimaging measures) | Pre-treatment assessment (week 2) and post-treatment assessment (week 6)
  The Neveu et al. (2018) task will be used, which consists of three phases: two rating phases and one decision phase with 50 food images. Participants have to answer on a 5-point Likert scale how healthy they consider the food to be (block 1) and how much they like the taste of the food (block 2). In the third block, the participant decides whether they prefer to eat a neutral reference food (calculated from the previous two blocks) or an alternative food. These forced choices lead to cognitive conflict when the reference food is considered tastier and the alternative food healthier or vice versa. Among trials with cognitive conflict, the choice of the healthier food is defined as a controlled choice, and the choice of the tastier food as an uncontrolled choice. Activation will be compared between the controlled vs. uncontrolled choice conditions.
  The task will be analysed to assess the brain activity associated with the task, using a psychophysiological interaction analyses (PPI).
Changes in Brain connectivity at rest (neuroimaging measures) | Pre-treatment assessment (week 2) and post-treatment assessment (week 6)
  Participants will be instructed to remain still, with their eyes closed, trying not to think about anything in particular for 9 minutes to obtain images to study the resting connectivity of different brain networks. On the one hand, an independent component analyses (ICA) will be performed, which will allow comparison of the different brain networks, as a whole, between the groups, with special interest in those that have been shown to be altered in the PD population. On the other hand, seed-based connectivity analyses will be performed, in which changes in functional connectivity between the CPFDL and the rest of the brain will be observed.
Changes in White matter integrity (neuroimaging measures) | Pre-treatment assessment (week 2) and post-treatment assessment (week 6)
  Participants will be asked to remain still for 10 minutes to obtain diffusion tensor imaging (DTI) which provides indirect measurements of the architecture and connectivity of white matter fibres. The study of the DTI images will be carried out with the FSL programme, which allows the integrity of the white matter of the different groups to be measured by evaluating the fractional anisotropy (FA) and apparent diffusion coefficient (ADC) maps.
Waist-to-height ratio (WHtR). Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  To take these measurements at home, participants should ask someone for help and follow our instructions. WHtR results from WC divided by the height measured standing with heels close together and trunk erect.
Food Craving. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Change in Food Craving. Food Craving Questionnaire State-reduced (FCQ-S-r)consists of 15 items to be scored on a 5-point scale ranging from strongly disagree to strongly agree. A higher score indicates higher state of craving at the time of the assessment
Eating behaviour. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Diet information during the last year (pre-treatment), two last weeks (post-treatment) and 3 last months (follow-up) will be collected through a 52-item Food frequency questionnaire (CFA). Participants must record quantities of all the foods and drinks consumed during those periods. Data are transformed into total calories and calories from fats, carbohydrates, and sugars
Physical activity behaviour. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  International Physical Activity Questionnaire (IPAQ; www.ipaq.ki.se): is a questionnaire with 7 questions on physical activity during the last week, as well as walking and sitting time.It evaluates physical activity related to work, activity at home and free time determines the degrees of activity based on the metabolic equivalents (MET) consumed.Higher scores indicate greater physical activity
Exercise adherence. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The following question will be asked using a visual analogue scale (VAS): In the last 2 weeks or 3 months, to what extent did you follow the exercise guidelines given to you by the programme's physical trainer? (0 = I did not follow the exercise recommendations at all; 100 = I absolutely followed the exercise recommendations).
Adherence to diet. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The following question will be asked using a visual analogue scale (VAS): In the last 2 weeks or 3 months, how well did you follow the dietary guidelines given by the nutritionist in the programme (0 = I did not follow the diet at all; 100 = I followed the diet absolutely).
Depression symptoms. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Beck Depression Inventory will be administered to test depression symptoms.The scores range from 0 to 63 points. The higher the score, the greater the severity of depressive symptoms
Anxiety and Stress. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Depression Anxiety Stress Scale-21 (DASS-21) will be used, taking into account scores on the stress and anxiety subscales. The scores for both subscales range from 0 to 21, a higher score indicating higher anxiety or stress
Non homeostatic eating. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Dutch Eating Behaviour Questionnaire (DEBQ) will be administered to assess restrictive eating behaviours related to external cues and emotional states. Higher scores in each subscale reflect higher level of restrained, emotional, and external eating, respectively.The DEBQ uses a 5-point Likert scale, ranging from never (1) to very often (5). The average score is calculated for each subscale by adding scores obtained from individual items and dividing them by the number of items included in a subscale (mean range: 1-5).
Reward-related eating. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Reward-Based Eating Scale (RED) is a 13 items questionnaire that evaluates worries about foods, losing intake control and absence of satiety. Higher scores reflect higher reward-based eating drive.
Emotional eating. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Coping subscale of the Palatable Eating Motives Scale (PEMS) will be used to evaluate the intentionality for eating palatable foods to face negative emotions. The coping subscale includes items that are scored on a 5-point Likert-type scale, the total range being from 5 to 25 points. Low scores indicate that the person rarely resorts to the consumption of pleasant foods as a strategy to cope with negative emotions or stressful situations. High scores suggest that the person frequently uses palatable food as a strategy to cope with stress or negative emotions, which may be related to unhealthy eating habits or emotional eating patterns.
Emotion Regulation Strategies. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Emotion Questionnaire (ERQ) consists of 10 items to examine cognitive reappraisal and expressive suppression strategies. In cognitive reappraisal the highest score (42) is associated with better emotional outcomes while in expressive suppression the highest score (28) is linked to poorer well-being. Each item is rated on a Likert scale from strongly disagree (1) to strongly agree (7).
Motor inhibition. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Motor inhibition will be assessed using FoodT. In the FoodT app reaction time for the high-calorie and low-calorie foods paired with the go and the no-go signal. The average response time for go and no-go items will be calculated according to the type of images (appetizing and healthy foods), and commission errors will be recorded.
Cognitive inhibition. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Using a Stroop task with food, the interference of food-related words on task performance can be measured as an assessment of cognitive inhibition.
Delay of gratification. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Score on the Food Delay Discounting will be used to measure the sensitivity to immediate rewards vs higher value rewards delayed. The participant's choices are recorded for each trial. Each trial varies in terms of the amount of reward and the amount of time to wait. To model the decisions, a hyperbolic discounting function is generally used.
Inhibition and activation systems. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  This will be assessed using the Punishment Sensitivity and Reward Sensitivity Questionnaire (PSRSQ) of 48 items. Responses in the scale are in a "yes/no" format. Higher punishment sensitivity scores are associated with lower number of punishable errors while higher reward sensitivity scores are linked to higher number of passive avoidance errors.
Self-reported impulsivity. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Self-reported impulsivity will be measured with Impulsive behaviour scale (UPPS-P). It consists of 20 items scored on a four point Likert scale, ranging from strongly agree (1) to strongly disagree (4). Higher scores mean worse outcome in impulsivity, while lower scores are related to better self-control and regulation
Working Memory. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Working Memory will be assessed using N-back Task score based on accuracy and reaction times. Higher accuracy scores indicate stronger working memory and attention, while faster reaction times are linked to quicker processing speed and decision-making.
Cognitive flexibility. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Wisconsin Card Sorting Test will be administered to measure shift strategy in response to changing contingencies. There are128 trials where more correct responses, fewer perseverative and non perseverative errors, and more completed categories (max 6) are related to better performance
Decision making. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Iowa Gambling Task will be used to assess decision-making using money rewards.

OTHER OUTCOMES:
Descriptive measures | Pre-treatment assessment (week 2)
  A socio-demographic questionnaire will be administered to examine age, education, gender, socio-economic variables and clinical variables to consider exclusion and inclusion criteria. All these variables are qualitative.
Depression Symptoms. Screening | Pre-treatment assessment (week 2)
  The Beck Depression Inventory (BDI-II) will also be used to rule out major depressive symptoms as an exclusion criteria. The scores range from 0 to 63 points. Participants with a score higher than 29, indicative of severe symptoms, will be excluded.
Anxiety Symptoms. Screening | Pre-treatment assessment (week 2)
  The anxiety subscale of the DASS-21 will also be used to rule out symptoms of major anxiety as an exclusion criterion. The scores for both subscales range from 0 to 21. Participants with a score higher than 8, indicative of severe symptoms, will be excluded from the study.
Eating and Weight Patterns. Screening | Pre-treatment assessment (week 2)
  Questionnaire on Eating and Weight Patterns-5 (QEWP-5) is adapted to DSM-5 criteria and will be used to exclude people with binge eating problems and bulimia. The QEWP-5 is not scored on a traditional numerical scale like other psychological tests; instead, responses are used to identify the presence of eating disorder symptoms. Positive responses to key questions about the frequency of binge eating, compensatory behaviors, and emotional distress may indicate the presence of an eating disorder.
Using of Health Resources | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Health Resources Questionnaire asks how often and why people have needed medical care and medicines in the last 3 month to measure the impact of the intervention in terms of health uses. Fewer visits to health professionals will be indicative of improvement.
Motivation to change | Pre-treatment assessment (week 2)
  Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) adapted to excess weight will be used to assess motivation to change habits. It has 18 items that score readiness to change in people with abusive food use with a five point Likert scale, ranging from strongly disagree (1) to strongly agree (5). Higher scores mean better outcome in relation to motivation to change, while higher scores on ambivalence suggest doubts about the motivation to change.
Stigma | Pre-treatment assessment (week 2)
  A yes/no question will be asked to record whether or not participants have experienced weight stigma in the past and a VAS scale from 0 to 100 where they can rate the degree to which they have experienced stigma.
Previous treatment history | Pre-treatment assessment (week 2)
  History of previous treatment, from pharmacological or nutritional to psychological, should be recorded.
Hormone levels (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine hormone levels (pg/ml) of estradiol, progesterone, cortisol, leptin, adiponectin, TSH, thyroxine, triiodothyronine, ghrelin, glucagon and GLP-1. A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Glucose and triglycerides levels (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will glucose and triglycerides levels (mg/dl). A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Insulin levels (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine concentration of insulin (U/ml). A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Inflammatory parameters (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine concentration of IL-6 (pg/ml), CRP (mg/L) and TNF-alpha (pg/ml). In addition, genetic analyses will be performed by sequencing candidate genes. A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Satiety markers (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine PYY (3-36) levels (pg/ml). A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Genetic analyses (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Fasting blood tests will determine genetic analyses will be performed by sequencing candidate genes. Genome-wide association analysis is proposed to identify new genes and variants associated with PD such as ZFP36, GAD2 on chromosome 10p12, Neuromedin β with whole exome sequencing and methylation analysis.A total of 10 ml of blood will be collected and centrifuged to separate the plasma from the rest and stored at -80ºC
Oral microbiota (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Saliva sample tests will determine oral microbiota (microbial taxa). It will be collected using three swabs (right cheek, left cheek, tongue) that will be stored at -80ºC
Gut microbiota (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project.
  Participants will collect fecal samples and 1.5 g of the top layer will be stored in tubes at -80ºC. Testing of faecal samples will determine gut microbiota composition (microbial taxa).
Proteomics analysis. (Biological samples collection) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Biological samples will be collected and deep-frozen in the CIMCYC until mass analyses are performed at the end of the project. Proteomics analyses will determine concentration of proteins (mg/mL).
  Samples will be collected in plastic bottles, centrifuged and stored at -80ºC
Quality of Life (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The SF-36 (Short Form 36 Health Survey) is one of the most widely used questionnaires to measure health-related quality of life.
  It consists of 36 questions assessing eight key dimensions: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role and mental health. Each dimension is scored on a scale of 0 to 100, where 0 represents the worst health status and 100 the best.
Years of Life Adjusted for Quality (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Years of Life Adjusted for Quality (QALY) is a measure used in healthcare to assess the value of medical treatments or interventions, combining quantity and quality of life. One QALY is equivalent to one year of life in full health. If a person lives a year with a reduced quality of life (due to illness, for example), a value of less than 1 is assigned, depending on the degree of well-being. This metric allows the effectiveness of different interventions to be compared, helping in health decision-making and resource allocation. It combines life years and quality (from SF-36) used in economic evaluation and cost-utility analyses of the intervention
BMI (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The BMI will be used to assess the success of the intervention in the cost-effectiveness calculations.
Intensity of Food Craving (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The FCQ-S-r will be used to assess the success of the intervention in the cost-effectiveness calculations.
Health Resource Costs (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Health Resource Questionnaire will be used to assess the success of the intervention in the cost-effectiveness calculations.
iTBS Session Staff Time (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Cost of a Clinical Psychology Area Specialist (FEA) for 3 minutes per session over 10 days, based on Andalusian Health Service remuneration will be used to assess the success of the intervention in the cost-effectiveness calculations.
Inhibitory Control Training Session Staff Time (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Cost of a Clinical Psychology Area Specialist (FEA) for 10 minutes per session over 10 days, based on Andalusian Health Service remuneration will be used to assess the success of the intervention in the cost-effectiveness calculations.
Equipment Costs (Measures to calculate cost effectiveness, cost utility and budget impact analyses) | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Cost of fMRI and iTBS equipment will be used to assess the success of the intervention in the cost-effectiveness calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vilar López, Ph.D., Principal Investigator — Universidad de Granada
Locations (1):
- Mind, Brain and Behavior Research Center at University of Granada (CIMCYCUGR), Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee and who provide a methodologically sound proposal. Proposals should be directed to rvilar@ugr.es

REFERENCES:
- See also: Project website — http://trainep.ugr.es/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT06668077/Prot_SAP_002.pdf
  • Informed Consent Form (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT06668077/ICF_001.pdf